CLINICAL TRIAL: NCT05761704
Title: A Prospective Exploratory Clinical Observation of Two Short-term Regimens (Dual Antiplatelet or Novel Oral Anticoagulant) for Subjects With Non-valvular Atrial Fibrillation After Left Atrial Appendage Occlusion by LAMax LAAC® Device
Brief Title: Exploratory Observation of Two Short-term Regimens After LAA Occlusion by LAMax LAAC® Device for Subjects With Non-valvular Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAHZJU CT021
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Atrial Fibrillation; Left Atrial Appendage Closure; Ischemic Stroke; Device-related Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual antiplatelet (Experimental): Aspirin 100 mg + clopidogrel 75 mg for 4 weeks post-LAAC; followed by aspirin/clopidogrel for 4-24 weeks post-LAAC; recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).
  Interventions: Drug: Dual antiplatelet
- Novel oral anticoagulant (Experimental): Conventional dose NOAC for 4 weeks post-LAAC; followed by aspirin/clopidogrel for 4-24 weeks post-LAAC; recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).
  Interventions: Drug: Novel oral anticoagulant

INTERVENTIONS:
Drug: Dual antiplatelet — Aspirin 100 mg + clopidogrel 75 mg for 4 weeks post-LAAC; followed by aspirin/clopidogrel for 4-24 weeks post-LAAC; recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).
  Arms: Dual antiplatelet
Drug: Novel oral anticoagulant — Conventional dose NOAC for 4 weeks post-LAAC; followed by aspirin/clopidogrel for 4-24 weeks post-LAAC; recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).
  Arms: Novel oral anticoagulant

SUMMARY:
This is a prospective, single-center, randomized, exploratory clinical observation to explore the overall benefit of short-term dual antiplatelet or novel oral anticoagulant regimens after left atrial appendage (LAA) occlusion by LAMax LAAC® occluder for subjects with non-valvular atrial fibrillation (AF), which will provide a basis for subsequent research on real-world safety and efficacy of LAA closure (LAAC).

DETAILED DESCRIPTION:
Anticoagulation is necessary after transcatheter left atrial appendage closure (LAAC) and is important to prevent thrombosis and device-related thrombosis (DRT). Bleeding events and stroke should be reduced while reducing thrombosis. Based on the characteristics of the LAMax LAAC® device, experts recommend studying short-term medication regimens for patients with non-valvular atrial fibrillation after LAAC. This trial is a prospective, single-center, randomized, open-label and parallel design. It is estimated that 54 patients will take part in the study. Subjects with non-valvular atrial fibrillation undergo transcatheter LAAC using the LAMax LAAC® device, and then are randomly enrolled in observation group 1/observation group 2 of the medication regimen in a 1:1 ratio after LAAC.

Observation group 1 (dual antiplatelet group, 27 subjects): 4 weeks post-LAAC (aspirin 100 mg + clopidogrel 75 mg); 4-24 weeks post-LAAC (aspirin/clopidogrel); recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).

Observation group 2 (novel oral anticoagulant group, 27 subjects): 4 weeks post-LAAC (conventional dose NOAC); 4-24 weeks post-LAAC (aspirin/clopidogrel); recommended long-term aspirin treatment after 24 weeks (clopidogrel can be used instead if aspirin is intolerant).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients ≥ 18 years old with non-valvular atrial fibrillation (AF);
* 2. Subjects with LAAC indications: according to the 2023 SCAI/HRS Expert Consensus Statement on Transcatheter Left Atrial Attachment Closure, transcatheter LAAC is suitable for non-valvular AF patients with high risk of thromboembolism but unsuitable for long-term use of oral anticoagulants (OACs), including the following situations:

  1. Have a much higher risk of having stroke (CHA2DS2-VASc score: male ≥ 2 points, female ≥ 3 points),
  2. Have OAC intolerance or a much higher risk of bleeding (such as HAS-BLED score ≥ 3 points),
  3. Have sufficient life expectancy (minimum>1 year) and expected to improve quality of life after LAAC;
* 3. Successful left atrial appendage occlusion with LAMax LAAC® device;
* 4. Patients and their families fully understand the purpose of the study, voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* 1. Combined with other diseases except AF requiring long-term warfarin or other anticoagulant therapy;
* 2. Absolute contraindications for anticoagulation therapy or unacceptable bleeding risk with dual antiplatelet therapy;
* 3. Indications to dual antiplatelet therapy other than atrial fibrillation and/or left atrial appendage occlusion at the time of enrollment or predicted appearance of such indications within the duration of the trial (e.g. planned coronary revascularization);
* 4. Occluder dislocation, pericardial effusion (including new pericardial effusion and significantly increased pre-existing pericardial effusion) and other bleeding complications within 24 hours after LAAC;
* 5. Patients scheduled for catheter ablation after left atrial appendage electrical isolation and during the study;
* 6. Patients resistant to clopidogrel;
* 7. Patients requiring elective cardiac surgery;
* 8. Heart failure NYHA grade IV and not been corrected yet;
* 9. Patients with AF caused by rheumatic valvular heart disease, degenerative valvular heart disease, congenital valvular heart disease, severe mitral stenosis, aortic stenosis and other valvular diseases;
* 10. Initial atrial fibrillation, paroxysmal atrial fibrillation with a clear cause such as coronary artery bypass grafting (CABG) < 12 months, hyperthyroidism, etc.
* 11. Patients with acute myocardial infarction or unstable angina pectoris, or recent myocardial infarction < 12 months;
* 12. Patients with active bleeding, bleeding constitution or bleeding disorders, coagulation history and unhealed gastrointestinal ulcer;
* 13. Infective endocarditis, vegetation or other infections causing bacteremia, sepsis;
* 14. Female patients who are pregnant, lactating, or planning to become pregnant during this study;
* 15. Patients who have participated in other drug or device clinical trials and have not reached the endpoint;
* 16. Patients with renal insufficiency (endogenous creatinine clearance < 30ml/min) (using the standard Crockcroft-Gault formula) and/or advanced renal disease requiring dialysis;
* 17. Severe hepatic dysfunction (AST/ALT greater than 5 times the upper limit of normal or total bilirubin greater than 2 times the upper limit of normal);
* 18. Patients considered unsuitable for this study by the investigator.
* 19. Left atrial appendage has been removed, post heart transplantation, post atrial septal repair, or post occluder implantation;
* 20. Post prosthetic heart valve replacement;
* 21. Allergic to or contraindication to metal nickel alloy, aspirin, clopidogrel, contrast agent, heparin and other anticoagulants, etc;
* 22. Patients who have placed other instruments in the cardiovascular cavity and are unable to place the LAA occluder;
* 23. LVEF（left ventricular ejection fraction, by Simpson method）<35%；
* 24. Clear thrombus is found in the heart before LAAC;
* 25. TEE examination: the maximal orifice diameter of LAA is less than 12 mm, or more than 36 mm;
* 26. Residual flow after LAAC >5mm；
* 27. Patent foramen ovale with high risk;
* 28. Mitral stenosis with a valve area <1.5cm2;
* 29. Left atrial diameter (antero-posterior diameter) > 65mm, or pericardial effusion more than a small amount, the depth of local effusion > 10 mm;
* 30. Contraindications to X-ray, or not suitable for TEE examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related thrombosis | 24 weeks post-LAAC
  Incidence of device-related thrombosis (DRT) at the visit of 4 weeks post-LAAC documented by CTA and the visit of 24 weeks post-LAAC documented by transesophageal echocardiogram (TEE).
Incidence of stroke and transient ischemic attack | 24 weeks post-LAAC
  Incidence of stroke (classified as ischemic, hemorrhagic, or unspecified) and transient ischemic attack (TIA) before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.

SECONDARY OUTCOMES:
Incidence of bleeding events | 24 weeks post-LAAC
  Incidence of bleeding events before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.
Incidence of systemic embolic events | 24 weeks post-LAAC
  Incidence of systemic embolic events before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.
Incidence of procedure-related complications | 24 weeks post-LAAC
  Incidence of procedure-related complications (including device embolization, significant pericardial effusion) before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.
Incidence of composite clinical endpoint events | 24 weeks post-LAAC
  Incidence of composite clinical endpoint events (including death, myocardial infarction, stroke, TIA) before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.
Incidence of all-cause mortality | 24 weeks post-LAAC
  Incidence of all-cause mortality (including cardiac death, non-cardiac death, and unexplained death) before discharge or at 7 days, 4 weeks, and 24 weeks post-LAAC.
Incidence of myocardial infarction | 24 weeks post-LAAC
  Incidence of myocardial infarction before discharge or at 7 days, 4 weeks and 24 weeks post-LAAC.
Incidence of major bleeding | 24 weeks post-LAAC
  Incidence of major bleeding (BARC type 3 and 5) before discharge or at 7 days, 4 weeks and 24 weeks post-LAAC.
Adverse events | 24 weeks post-LAAC
  Adverse events on the day of surgery, before discharge, or at 7 days, 4 weeks, and 24 weeks post-LAAC.

CONTACTS AND LOCATIONS:
Overall Officials: Youqi Fan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China